CLINICAL TRIAL: NCT03296345
Title: Adjuvant Low-dose Ketamine in Pediatric Sickle Cell Vaso-occlusive Crisis (AKTSS)
Brief Title: Adjuvant Low-dose Ketamine in Pediatric Sickle Cell Vaso-occlusive Crisis
Acronym: AKTSS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-010
Record Dates: First submitted 2017-01-09; First posted 2017-09-28 (Actual); Results first posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-03

CONDITIONS: Sickle Cell Disease; Vaso-Occlusive Crisis
Keywords: Ketamine; Sickle Cell Disease; Vaso-Occlusive Episode
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Active Comparator): Prior to the second dose of IV opiates, the experiment was to give patients a single IV bolus of ketamine at the dose of 0.2 mg/kg. Pain scores were collected using the FACES scale currently in place. In consenting patients, chart review was performed with the following data collected: mg/kg/hour of morphine equivalents, pain scores on admission, during the encounter, and at discharge, the time to 50% pain reduction, and whether or not the patient was discharged.
  In addition, a survey, which is attached, was given to patients/families at the time of drug administration to determine if they experienced a subjective improvement in their pain and if they suffered any undue side effects due to drug administration.
  Interventions: Drug: Ketamine
- Historical Control (No Intervention): Patient data from at least one but up three patient encounters within the prior year were compared to their visit in which they were given adjuvant ketamine, using the outcome measures in the "Intervention" arm. Since this a historical control study, patients acted as their own controls in the above manner. Patients were allowed to re-enroll 4 weeks after presentation, which is typically considered a separate vaso-occlusive episode in the literature.

INTERVENTIONS:
Drug: Ketamine — The intervention is IV low-dose bolus ketamine as an adjuvant to standard therapy (IV opiates and NSAIDs).
  Other Names: Ketalar
  Arms: Intervention

SUMMARY:
Acute vaso-occlusive episodes (VOEs) in sickle cell disease (SCD) are primarily managed with opioids. Tolerance and hyperalgesia to opioids develops due to N-methyl-D-aspartate (NMDA)-receptor mediated activation of the nociceptive system, and as a receptor antagonist, ketamine mitigates this. Intravenous (IV) ketamine has demonstrated efficacy in reducing post-operative, chronic, and cancer-related pain in pediatrics, as well as in reducing time to pain control in the emergency department (ED) in adults. Limited studies suggest efficacy in adult opioid-refractory SCD patients. This study is investigating the safety and tolerability of adjuvant low-dose IV ketamine bolus for pediatric SCD VOE in the ED, as well as its efficacy in improving pain control and reducing hospitalization.

DETAILED DESCRIPTION:
In this cohort study, all consenting pediatric sickle-cell patients between 10 and 25 years old who were cared for at UCSF Benioff Children's Hospital Oakland (UCSFBCHO) presenting to the emergency department for VOC were enrolled in the study. Patients were compared to themselves in a time series, pre and post exposure to the study intervention (low-dose ketamine bolus at 0.2 mg/kg x 1 prior to second dose of IV opiate). The pediatric FACES pain scale was used to measure pain scales at pre-designated time points in the ED per standard nursing protocol (FACES for younger kids, visual analog scale in adolescents/young adults). Opiate usage was summed in the ED, converted to mg/kg/hour of morphine equivalents (since different opioids agents were given to different patients based on individual historical efficacy, and since length of stay in the emergency room could affect total morphine equivalents received), and compared between the pre and post-intervention groups. In addition, length of stay, time to 50% pain control, presentation and discharge pain scores, and likelihood of discharge from the ED were compared. Data was be collected via chart review in the UCSFBCHO system by study investigators. Pre-intervention data from the past three patient encounters (e.g., the mean of the mg/kg/hour of morphine equivalents used in the last three patient encounters prior to receipt of ketamine) was compared to the post intervention data. In addition, a survey, which is attached, was given to patients/families at the time of the drug administration to attempt to discern if patients subjectively experienced improvement in their pain and if they experienced any negative side effects due to the drug administration. Monitoring for adverse events was recorded for each patient encounter.

ELIGIBILITY:
Inclusion Criteria:

* All English-speaking, sickle cell patients who receive their care at UCSFBCHO in the Department of Hematology who are 8-to-25-years-old presenting to the emergency department for VOC were asked to enroll.

Exclusion Criteria:

* Prior adverse reaction to ketamine
* Patients were asked during the consent process if they have ever received ketamine, and if so, if they had any serious adverse reaction, such as difficulty breathing, dysphoria, hallucinations, or allergic reaction. If they have, ketamine was not given to these patients.
* Patients who have received ketamine and experienced nausea or vomiting will be asked if they wish to receive the medication. If they do not, they did not receive ketamine.

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2016-06; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan B Cooper-Sood, MD, Principal Investigator — Children's Hospital and Research Center of Oakland
Locations (1):
- UCSF Benioff Children's Hospital and Research Center Oakland, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neri CM, Pestieau SR, Darbari DS. Low-dose ketamine as a potential adjuvant therapy for painful vaso-occlusive crises in sickle cell disease. Paediatr Anaesth. 2013 Aug;23(8):684-9. doi: 10.1111/pan.12172. Epub 2013 Apr 9. PMID 23565738
- [Background] Tawfic QA, Faris AS, Eipe N. Sickle cell pain management: are we missing the role of pronociception and neuropathic pain? Paediatr Anaesth. 2013 Nov;23(11):1104-5. doi: 10.1111/pan.12269. No abstract available. PMID 24088202
- [Background] Jennings CA, Bobb BT, Noreika DM, Coyne PJ. Oral ketamine for sickle cell crisis pain refractory to opioids. J Pain Palliat Care Pharmacother. 2013 Jun;27(2):150-4. doi: 10.3109/15360288.2013.788599. Epub 2013 May 21. PMID 23692261
- [Background] Zempsky WT, Loiselle KA, Corsi JM, Hagstrom JN. Use of low-dose ketamine infusion for pediatric patients with sickle cell disease-related pain: a case series. Clin J Pain. 2010 Feb;26(2):163-7. doi: 10.1097/AJP.0b013e3181b511ab. PMID 20090444
- [Background] Riha H, Aaronson P, Schmidt A. Evaluation of analgesic effects of ketamine through sub-dissociative dosing in the ED. Am J Emerg Med. 2015 Jun;33(6):847-9. doi: 10.1016/j.ajem.2015.03.045. Epub 2015 Mar 25. No abstract available. PMID 25865160
- [Background] Beaudoin FL, Lin C, Guan W, Merchant RC. Low-dose ketamine improves pain relief in patients receiving intravenous opioids for acute pain in the emergency department: results of a randomized, double-blind, clinical trial. Acad Emerg Med. 2014 Nov;21(11):1193-202. doi: 10.1111/acem.12510. PMID 25377395
- [Background] Drake AB, Milne WK, Carpenter CR. Hot Off the Press: Subdissociative-dose Ketamine for Acute Pain in the Emergency Department. Acad Emerg Med. 2015 Jul;22(7):887-9. doi: 10.1111/acem.12705. Epub 2015 Jun 30. No abstract available. PMID 26130219
- [Background] Miller JP, Schauer SG, Ganem VJ, Bebarta VS. Low-dose ketamine vs morphine for acute pain in the ED: a randomized controlled trial. Am J Emerg Med. 2015 Mar;33(3):402-8. doi: 10.1016/j.ajem.2014.12.058. Epub 2015 Jan 7. PMID 25624076
- [Background] Uprety D, Baber A, Foy M. Ketamine infusion for sickle cell pain crisis refractory to opioids: a case report and review of literature. Ann Hematol. 2014 May;93(5):769-71. doi: 10.1007/s00277-013-1954-3. Epub 2013 Nov 15. PMID 24232306
- [Background] Tawfic QA, Faris AS, Kausalya R. The role of a low-dose ketamine-midazolam regimen in the management of severe painful crisis in patients with sickle cell disease. J Pain Symptom Manage. 2014 Feb;47(2):334-40. doi: 10.1016/j.jpainsymman.2013.03.012. Epub 2013 Jul 12. PMID 23856095
- [Background] Ahern TL, Herring AA, Anderson ES, Madia VA, Fahimi J, Frazee BW. The first 500: initial experience with widespread use of low-dose ketamine for acute pain management in the ED. Am J Emerg Med. 2015 Feb;33(2):197-201. doi: 10.1016/j.ajem.2014.11.010. Epub 2014 Nov 15. PMID 25488336

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Participants: Intervention: Prior to the second dose of IV opiates, the experiment was to give patients a single IV bolus of ketamine at the dose of 0.2 mg/kg.
  Ketamine: The intervention was IV low-dose bolus ketamine as an adjuvant to standard therapy (IV opiates and NSAIDs).
  Ultimately, 62 patient encounters were enrolled in the study.
  Historical Control: Patient data from at least one but up three patient encounters within the prior year were compared to their visit in which they were given adjuvant ketamine, using the outcome measures in the "Intervention" arm. Since this a historical control study, patients acted as their own controls in the above manner. Patients were allowed to re-enroll 4 weeks after presentation, which is typically considered a separate vaso-occlusive episode in the literature.
Period: Overall Study
Arm/Group | Study Participants
Started | 62
Completed | 62
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Participants: Intervention: Prior to the second dose of IV opiates, the experiment was to give patients a single IV bolus of ketamine at the dose of 0.2 mg/kg.
  Ketamine: The intervention is IV low-dose bolus ketamine as an adjuvant to standard therapy (IV opiates and NSAIDs).
Arm/Group | Study Participants
Number analyzed (Participants) | 62
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 18.1 [14 to 24]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 61
  White | 0
  More than one race | 0
  Unknown or Not Reported | 1
Site of pain on presentation [Number; unit: participants]
  Back | 22
  Extremity | 16
  Chest | 12
  Whole body | 5
  Abdomen | 4
  Other | 3
  Unknown | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events [Safety and Tolerability]
Description: The number of serious and minor adverse events was measured via patient-completed survey as well as by nurse and medical providers on presentation to the emergency department (ED). Serious adverse events are defined as cardiorespiratory events requiring intervention. Minor adverse events are defined as nausea/vomiting, emergence reaction (dysphoria; hallucinations; frightening dreams), and a sense of de-realization or "dreamy" sensation. Both study providers and patients themselves, via a survey that the parent and/or patient (based on age) fills out post receipt of ketamine, reported serious and minor adverse events.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: Prior to the second dose of IV opiates, the experiment was to give patients a single IV bolus of ketamine at the dose of 0.2 mg/kg.
  Ketamine: The intervention was IV low-dose bolus ketamine as an adjuvant to standard therapy (IV opiates and NSAIDs).
  Ultimately, 62 patient encounters were enrolled in the study.
Arm/Group | Intervention
Number analyzed (Participants) | 62
Participants
  Serious adverse events | 0
  Nausea/vomiting | 4
  Emergence of emergence-like symptoms | 4
  Dream-like/de-realized sensation | 26
  Blurry vision | 3
  Dizziness | 2
  Floating sensation | 1
  Heavy sensation | 1
  Dry mouth | 1
  No adverse event | 20

2. Secondary Outcome: Effect of Low-dose Ketamine (LDK) on Opioid Usage in the ED
Description: Opioid usage for at least one but up to three prior patient visits in the last one year for each patient enrolled in the study was summarized, expressed as morphine equivalents in mg/kg/h, to account for different types of opioids used per patient preference, and then this was compared to the intervention group that received LDK. Percent change in opioid usage (expressed as morphine equivalents in mg/kg/h) is reported).
Time Frame: Up to one year prior and after LDK administration on day 1 of the study in the ED
Population: 62 enrolled patient-encounters were compared to their prior visits individually. At least one but up to three prior visits were averaged and compared to the intervention visit.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Intervention
Number analyzed (Participants) | 62
percent change | -15 [-28 to -2.3]
Statistical Analysis 1: Comparison: Intervention; Test type: Other; p = 0.004, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -15, 95% CI 2-sided [-28 to -2.3]

3. Secondary Outcome: Effect of Low-dose Ketamine on Pain Scores on Presentation to the ED
Description: Patient pain scores at presentation for the enrolled encounters and for at least one but up to three visits prior to receipt of ketamine in the last one year, were assessed. At least one but up to three prior visits were averaged and compared to the intervention visit. Pain was assessed using the faces pain scale which consists of a series of line diagrams of faces with expressions of increasing distress. The score ranges from 0 (no pain) to 10 (the worst pain).
Time Frame: Up to one year prior and on presentation to the ED after LDK administration
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Intervention | Historical Control
Number analyzed (Participants) | 62 | 62
Score on a scale | 9.23 [8.98 to 9.47] | 9.08 [8.83 to 9.34]
Statistical Analysis 1: Comparison: Intervention vs Historical Control; Test type: Other; p = 0.38, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Effect of Low-dose Ketamine on Discharge Rates From the ED
Description: Percent discharge from the ED for intervention group and for at least one but up to three visits prior to receipt of ketamine in the last one year, were assessed. Participants were assigned a "0" if discharged or "1" if not discharged.
Time Frame: Up to one year prior to receipt of ketamine for the historical control arm/group and up to 18 months for the intervention arm/group
Measure: Number; unit: percentage of participants
Arm/Group | Intervention | Historical Control
Number analyzed (Participants) | 62 | 62
percentage of participants | 33 | 17
Statistical Analysis 1: Comparison: Intervention vs Historical Control; Test type: Other; p = 0.58, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Subjective Effect of Low Dose Ketamine on Pain Relief Assessed Via a Patient Survey
Description: After receipt of LDK, patients and/or their parents, based on age, filled out a survey based on a Likert scale regarding their agreement (Strongly Disagree to Strongly Agree) with the following statements: Achieved faster pain relief with LDK, Achieved more complete pain relief with LDK, and Desire to receive LDK in a future vaso-occlusive crisis. There is also an area where patients could provide general comments regarding their experience in receiving LDK.
  Count of Participants who agree or strongly agree for each question are reported.
Time Frame: after LDK administration on day 1 of the study in the ED
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 62
Participants
  Achieved faster pain relief? | 43
  Achieved more complete pain relief? | 30
  Desire to receive LDK in the future? | 49

6. Secondary Outcome: Effect of Low-dose Ketamine on Patient Pain Scores on Discharge From the ED/Admission to the Hospital
Description: Patient pain scores at time of discharge from the ED/admission to the hospital for at least one but up to three visits prior to receipt of ketamine in the last one year, were assessed. At least one but up to three prior visits were averaged and compared to the intervention visit. Pain scores post receipt of ketamine are presented for the intervention group. Pain was assessed using the faces pain scale which consists of a series of line diagrams of faces with expressions of increasing distress. The score ranges from 0 (no pain) to 10 (the worst pain).
Time Frame: At time of discharge from the ED/admission to the hospital (up to one year prior and after LDK administration)
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Intervention | Historical Control
Number analyzed (Participants) | 62 | 62
Score on a scale | 7.15 [6.61 to 7.68] | 7.26 [6.84 to 7.68]
Statistical Analysis 1: Comparison: Intervention vs Historical Control; Test type: Other — A Wilcoxon sign-rank, given non parametric data, was used to compare the intervention and historical control groups for statistical significance, while a student's t-test was used to estimate effect size; p = 0.76, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Effect of Low-dose Ketamine on Percent Difference of Length of Stay (LOS) in the ED
Description: Length of stay (LOS) in minutes in the ED for at least one but up to three visits prior to receipt of ketamine in the last one year, were assessed.
Time Frame: Up to one year prior to and after LDK administration on day 1 of the study in the ED
Measure: Mean (95% Confidence Interval); unit: LOS in minutes
Arm/Group | Intervention | Historical Control
Number analyzed (Participants) | 62 | 62
LOS in minutes | 273.5 [241.3 to 305.6] | 217.3 [200.0 to 234.5]

8. Secondary Outcome: Effect of Low-dose Ketamine on Time to 50% Pain Reduction
Description: Time to 50% pain reduction (pain reported 50% less than baseline) in minutes for at least one but up to three visits prior to receipt of ketamine in the last one year, were assessed as historical controls. Pain was assessed using the faces pain scale which consists of a series of line diagrams of faces with expressions of increasing distress. The score ranges from 0 (no pain) to 10 (the worst pain).
Time Frame: Up to one year prior to and after LDK administration on day 1 of the study in the ED
Population: 16 participants reported a 50% pain reduction, and those 16 participants were included in the analysis of time to 50% pain reduction.
Measure: Mean (95% Confidence Interval); unit: time to 50% pain reduction in minutes
Groups:
- Historical Control: Patient data from at least one but up three patient encounters within the prior year were compared to their visit in which they were given adjuvant ketamine, using the outcome measures in the "Intervention" arm. Since this a historical control study, patients acted as their own controls in the above manner.
Arm/Group | Intervention | Historical Control
Number analyzed (Participants) | 16 | 16
time to 50% pain reduction in minutes | 116.1 [111.6 to 220.6] | 167.3 [117.0 to 217.5]

ADVERSE EVENTS:
Time Frame: 18 months
Description: Serious adverse events were defined per protocol as reaction to intervention causing cardiorespiratory compromise requiring medical intervention.
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/62
Serious Adverse Events (participants affected / at risk) | 0/62
Other Adverse Events (participants affected / at risk) | 42/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=62)
Nausea/vomiting (Gastrointestinal disorders) | 4
Emergence of emergence-like symptoms (General disorders) | 4
Dream-like/de-realized sensation (General disorders) | 26
Blurry vision (Eye disorders) | 3
Dizziness (Vascular disorders) | 2
Floating sensation (General disorders) | 1
Heavy sensation (General disorders) | 1
Dry mouth (General disorders) | 1

LIMITATIONS AND CAVEATS:
Given the study design (non-blinded, non-randomized), the effect of LDK on opioid usage and other secondary outcomes cannot be definitively associated with LDK itself given the possibility of a placebo effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-28): https://cdn.clinicaltrials.gov/large-docs/45/NCT03296345/Prot_SAP_000.pdf